CLINICAL TRIAL: NCT01925209
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group, Dose-finding, Pivotal, Phase 2b/3 Study to Evaluate the Efficacy, Safety, and Tolerability of Intravenous BYM338 at 52 Weeks on Physical Function, Muscle Strength, and Mobility and Additional Long Term Safety up to 2 Years in Patients With Sporadic Inclusion Body Myositis
Brief Title: Efficacy and Safety of Bimagrumab/BYM338 at 52 Weeks on Physical Function, Muscle Strength, Mobility in sIBM Patients
Acronym: RESILIENT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBYM338B2203
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Sporadic Inclusion Body Myositis
Keywords: sporadic inclusion body myositis,; myositis,; muscle wasting,; controlled clinical trial,; randomized,; body mass,; muscle function,; strength,; performance,; physical function
MeSH Terms: conditions — Myositis, Inclusion Body; Myositis; Muscular Atrophy | interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BYM338/bimagrumab 10 mg/kg (Experimental): Participants received study medication with BYM338 at 10 mg/kg from Day 1 to Week 52 and up to Week 104, administered by intravenous (i.v.) infusion every 4 weeks.
  Interventions: Drug: BYM338/bimagrumab
- BYM338/bimagrumab 3 mg/kg (Experimental): Participants received study medication with BYM338 at 3 mg/kg from Day 1 to Week 52 and up to Week 104, administered by i.v. infusion every 4 weeks.
  Interventions: Drug: BYM338/bimagrumab
- BYM338/bimagrumab 1 mg/kg (Experimental): Participants received study medication with BYM338 at 1 mg/kg from Day 1 to Week 52 and up to Week 104, administered by i.v. infusion every 4 weeks.
  Interventions: Drug: BYM338/bimagrumab
- Placebo (Placebo Comparator): Participants received matching placebo to BYM338 from Day 1 to Week 52 and up to Week 104, administered by i.v. infusion every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BYM338/bimagrumab — BYM338, a 150 mg/mL concentrate for solution for i.v. infusion, was provided in colorless glass vials with a rubber stopper and aluminum flip-off caps.
  Arms: BYM338/bimagrumab 1 mg/kg; BYM338/bimagrumab 10 mg/kg; BYM338/bimagrumab 3 mg/kg
Drug: Placebo — Matching placebo to BYM338 was provided in colorless glass vials with a rubber stopper and aluminum flip-off caps.
  Arms: Placebo

SUMMARY:
This study evaluated the efficacy, safety and tolerability of multiple doses of bimagrumab/BYM338 vs placebo, when administered intravenously (i.v.), on physical function, muscle strength, and mobility in patients with sporadic inclusion body myositis (sIBM).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with sporadic inclusion body myositis;
* Must be able to walk (assistive aids allowed, including intermittent use of wheelchair);

Key Exclusion Criteria:

* Must not have other conditions that significantly limit ability to move around;
* Must not be using corticosteroids. Must not have used systemic corticosteroid (at daily dose >=10mg prednisone) for the past 3 months;
* Must meet cardiovascular requirements;
* Must not be pregnant or nursing;
* Must not have a chronic active infection (e.g., HIV, hepatitis B or C, tuberculosis, etc.);

Ages: 36 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2016-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (11):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
- Australia (3):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Cauldfield, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Paris, France
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Tokushima, Tokushima
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Wakayama, Wakayama
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leiden
- Novartis Investigative Site, Zurich, Switzerland
- United Kingdom (3):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Hanna MG, Badrising UA, Benveniste O, Lloyd TE, Needham M, Chinoy H, Aoki M, Machado PM, Liang C, Reardon KA, de Visser M, Ascherman DP, Barohn RJ, Dimachkie MM, Miller JAL, Kissel JT, Oskarsson B, Joyce NC, Van den Bergh P, Baets J, De Bleecker JL, Karam C, David WS, Mirabella M, Nations SP, Jung HH, Pegoraro E, Maggi L, Rodolico C, Filosto M, Shaibani AI, Sivakumar K, Goyal NA, Mori-Yoshimura M, Yamashita S, Suzuki N, Katsuno M, Murata K, Nodera H, Nishino I, Romano CD, Williams VSL, Vissing J, Auberson LZ, Wu M, de Vera A, Papanicolaou DA, Amato AA; RESILIENT Study Group. Safety and efficacy of intravenous bimagrumab in inclusion body myositis (RESILIENT): a randomised, double-blind, placebo-controlled phase 2b trial. Lancet Neurol. 2019 Sep;18(9):834-844. doi: 10.1016/S1474-4422(19)30200-5. PMID 31397289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized into one of the four treatment arms in a 1:1:1:1 ratio.
Pre-assignment Details: The study included 4 epochs: screening (up to 28 days pre-treatment), treatment (from day 1 up to 52 weeks), treatment maintenance (from week 52 up to 104 weeks) and follow-up (28 days after last dose administration).
Period: Treatment Epoch
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Started | 63 | 63 | 63 | 62
Full Analysis Set | 63 | 63 | 63 | 62
Completed | 54 | 55 | 56 | 57
Not Completed | 9 | 8 | 7 | 5
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3 | 3 | 2
Not completed — Adverse Event | 3 | 5 | 3 | 1
Period: Maintenance Treatment Epoch
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Started | 49 | 46 | 52 | 50
Completed | 49 | 45 | 50 | 48
Not Completed | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Follow-up
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Started | 57 | 61 | 56 | 58
Completed | 56 | 55 | 55 | 54
Not Completed | 1 | 6 | 1 | 4
Not completed — Adverse Event | 1 | 4 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Non-compliance with study treatment | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS), which included all randomized participants who had received at least one dose of study drug and had at least one post-baseline efficacy assessment, was analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo | Total
Number analyzed (Participants) | 63 | 63 | 63 | 62 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (7.93) | 66.5 (8.72) | 69.4 (7.91) | 68.4 (8.12) | 68.1 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 23 | 23 | 89
  Male | 41 | 42 | 40 | 39 | 162

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6 Minute Walking Distance (6MWD) Test at Week 52
Description: The 6MWD test measured the distance (in meters) that a participant walked in a 6 minute timeframe. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: The Full Analysis Set (FAS), which included all randomized participants who had received at least one dose of study drug and had at least one post-baseline efficacy assessment, was considered for the analysis. Only those participants from the FAS who had both baseline and week 52 6MWD measurements were analyzed.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 61 | 63 | 63 | 62
meters | 8.63 (10.934) | 9.63 (10.770) | -10.27 (10.718) | -8.96 (10.765)
Statistical Analysis 1: Comparison: BYM338/Bimagrumab 10 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.2210, mixed model repeated measures; Mean Difference (Net) = 17.59, 99% CI 2-sided [-19.63 to 54.80], Standard Error of Mean 14.331
Statistical Analysis 2: Comparison: BYM338/Bimagrumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.1909, mixed model repeated measure; Mean Difference (Net) = 18.59, 99% CI 2-sided [-18.21 to 55.40], Standard Error of Mean 14.176
Statistical Analysis 3: Comparison: BYM338/Bimagrumab 1 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.9263, mixed models repeated measures; Mean Difference (Net) = -1.31, 99% CI 2-sided [-37.97 to 35.36], Standard Error of Mean 14.121

2. Secondary Outcome: Estimated Within Treatment Group Lean Body Mass (LBM) Ratio at Week 52
Description: LBM was measured via dual energy x-ray absorptiometry (DXA) and calculated as (LBM at Week 52/LBM at baseline)*100 . A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: The Full Analysis Set (FAS), which included all randomized participants who had received at least one dose of study drug and had at least one post-baseline efficacy assessment, was considered for the analysis. Only those participants from the FAS who had both baseline and week 52 LBM measurements were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 62 | 61 | 63 | 61
Percentage | 102.8 [101.4 to 104.2] | 100.4 [99.1 to 101.8] | 98.3 [97.0 to 99.6] | 97.2 [95.9 to 98.5]

3. Secondary Outcome: Change From Baseline in Quadriceps Quantitative Muscle Testing (QMT) on the Right Side at Week 52
Description: Quadriceps muscle strength was measured by portable fixed dynamometry (PFD) on the right side. A negative change from baseline indicates deterioration.
Time Frame: Baseline, Week 52
Population: The Full Analysis Set (FAS), which included all randomized participants who had received at least one dose of study drug and had at least one post-baseline efficacy assessment, was considered for the analysis. Only those participants from the FAS who had both baseline and week 52 QMT measurements were analyzed.
Measure: Least Squares Mean (Standard Error); unit: newtons
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 60 | 63 | 63 | 61
newtons | -12.44 (6.021) | -20.36 (5.843) | -14.89 (5.828) | -16.48 (5.830)

4. Secondary Outcome: Change From Baseline in Sporadic Inclusion Body Myositis (sIBM) Functional Assessment (sIFA) Score at Week 52
Description: Self-reported physical function was assessed by a newly developed patient reported outcome named sporadic inclusion body myositis (sIBM) functional assessment (sIFA). The sIFA consists of 11 items scored on an 11 point numerical rating scale from 0 (no difficulty) to 10 (unable to do) across 3 domains: upper body functioning, lower body functioning and general functioning. Participants completed the assessment where the recall period was the past week prior to completing the patient reported outcome (PRO). The total score on the sIFA scale ranges from 0 (minimum) to 110 (maximum). Higher values represent a worse outcome. A positive change from baseline indicates deterioration.
Time Frame: Baseline, Week 52
Population: The Full Analysis Set (FAS), which included all randomized participants who had received at least one dose of study drug and had at least one post-baseline efficacy assessment, was considered for the analysis. Only those participants from the FAS who had both baseline and week 52 sIFA measurements were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 61 | 63 | 60 | 61
score on a scale | 1.74 (1.915) | 3.56 (1.876) | 6.12 (1.899) | 6.85 (1.895)

5. Secondary Outcome: Estimated Annual Number of Falls Per Patient Within Treatment Group
Description: Participants documented any fall occurrences in a paper diary during the study.
Time Frame: Week 52
Population: as for baseline characteristics
Measure: Number; unit: Annual number of falls per participant
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 63 | 63 | 63 | 62
Annual number of falls per participant | 4.33 | 4.02 | 4.70 | 5.13

6. Secondary Outcome: Change From Baseline in Short Physical Performance Battery (SPPB) Score at Week 52
Description: The SPPB evaluated lower extremities function by testing gait speed, ability to keep standing balance and time to rise from a chair five times. The sub-score for each test ranged from 0 to 4. The summary score, which was a summation of scores from the 3 tests, ranged from 0 to 12. An increase in score indicates improvement in physical performance. A negative change from baseline indicates deterioration.
Time Frame: Baseline, Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 62 | 63 | 63 | 62
score on a scale | 0.0 (0.24) | 0.0 (0.23) | -0.5 (0.23) | -0.5 (0.23)

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 21/63 | 11/63 | 18/63 | 20/62
Other Adverse Events (participants affected / at risk) | 63/63 | 63/63 | 63/63 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338/Bimagrumab 10 mg/kg (N=63) | BYM338/Bimagrumab 3 mg/kg (N=63) | BYM338/Bimagrumab 1 mg/kg (N=63) | Placebo (N=62)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 1 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
RETINAL ARTERY OCCLUSION (Eye disorders) | 0 | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 0 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 2
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 1 | 0
VOLVULUS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INJURY ASSOCIATED WITH DEVICE (General disorders) | 0 | 0 | 1 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ENDOTRACHEAL INTUBATION COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
EYE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
SPINAL CORD INJURY CERVICAL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 1 | 3
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 0 | 0 | 1
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 0 | 1 | 0
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 0 | 1
BLADDER MASS (Renal and urinary disorders) | 0 | 0 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 1 | 0 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338/Bimagrumab 10 mg/kg (N=63) | BYM338/Bimagrumab 3 mg/kg (N=63) | BYM338/Bimagrumab 1 mg/kg (N=63) | Placebo (N=62)
ANAEMIA (Blood and lymphatic system disorders) | 5 | 3 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 4 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 6 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 6 | 3 | 6 | 3
DIARRHOEA (Gastrointestinal disorders) | 32 | 28 | 20 | 11
DRY MOUTH (Gastrointestinal disorders) | 5 | 1 | 3 | 4
DYSPHAGIA (Gastrointestinal disorders) | 5 | 4 | 1 | 5
NAUSEA (Gastrointestinal disorders) | 11 | 4 | 9 | 5
VOMITING (Gastrointestinal disorders) | 4 | 1 | 2 | 3
ASTHENIA (General disorders) | 1 | 3 | 4 | 6
FATIGUE (General disorders) | 9 | 4 | 14 | 7
OEDEMA PERIPHERAL (General disorders) | 5 | 9 | 9 | 7
PYREXIA (General disorders) | 3 | 1 | 3 | 5
FOLLICULITIS (Infections and infestations) | 4 | 2 | 0 | 1
INFLUENZA (Infections and infestations) | 2 | 4 | 4 | 2
NASOPHARYNGITIS (Infections and infestations) | 6 | 11 | 9 | 6
RHINITIS (Infections and infestations) | 0 | 1 | 1 | 4
SINUSITIS (Infections and infestations) | 1 | 4 | 1 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 11 | 14 | 10
URINARY TRACT INFECTION (Infections and infestations) | 4 | 4 | 2 | 4
CONTUSION (Injury, poisoning and procedural complications) | 14 | 23 | 22 | 22
FALL (Injury, poisoning and procedural complications) | 47 | 55 | 54 | 52
FOOT FRACTURE (Injury, poisoning and procedural complications) | 3 | 3 | 4 | 4
HEAD INJURY (Injury, poisoning and procedural complications) | 4 | 4 | 3 | 3
INJURY (Injury, poisoning and procedural complications) | 4 | 0 | 7 | 3
JOINT INJURY (Injury, poisoning and procedural complications) | 5 | 3 | 6 | 5
LACERATION (Injury, poisoning and procedural complications) | 6 | 5 | 12 | 9
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 7 | 10 | 9 | 10
LIMB INJURY (Injury, poisoning and procedural complications) | 5 | 7 | 2 | 8
SKIN ABRASION (Injury, poisoning and procedural complications) | 14 | 14 | 14 | 17
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 3 | 5 | 1 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 3 | 5 | 4 | 0
VITAMIN D DECREASED (Investigations) | 4 | 2 | 3 | 1
WEIGHT DECREASED (Investigations) | 9 | 4 | 8 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 | 3 | 3 | 1
GOUT (Metabolism and nutrition disorders) | 3 | 0 | 4 | 2
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 | 4 | 2 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4 | 2 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 6 | 12 | 3 | 11
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 | 14 | 19 | 15
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 8 | 14 | 9
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 6
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 32 | 43 | 25 | 13
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 4
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 | 4 | 7 | 4
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 | 11 | 7 | 8
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 4 | 13 | 7
DIZZINESS (Nervous system disorders) | 6 | 10 | 6 | 8
DYSGEUSIA (Nervous system disorders) | 5 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 12 | 4 | 14 | 9
HYPOAESTHESIA (Nervous system disorders) | 2 | 1 | 3 | 5
MUSCLE CONTRACTIONS INVOLUNTARY (Nervous system disorders) | 3 | 6 | 0 | 2
PARAESTHESIA (Nervous system disorders) | 0 | 2 | 2 | 5
ANXIETY (Psychiatric disorders) | 4 | 2 | 1 | 2
DEPRESSED MOOD (Psychiatric disorders) | 4 | 1 | 0 | 1
DEPRESSION (Psychiatric disorders) | 4 | 1 | 5 | 0
INSOMNIA (Psychiatric disorders) | 5 | 0 | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4 | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 5 | 5
ACNE (Skin and subcutaneous tissue disorders) | 12 | 19 | 8 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 6 | 6 | 6 | 1
RASH (Skin and subcutaneous tissue disorders) | 13 | 8 | 9 | 8
ROSACEA (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
HAEMATOMA (Vascular disorders) | 1 | 2 | 7 | 2
HYPERTENSION (Vascular disorders) | 7 | 7 | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.